CLINICAL TRIAL: NCT06072391
Title: Investigating the Endocrine-metabolic-immunological Axis During the Female Menstrual Cycle by Functional Genomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bonn (Other)
Collaborators: University Hospital, Bonn (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Marie-Christine Simon, PhD MSc RD, Jun. Prof. Dr. Marie-Christine Simon, University of Bonn
Other Study IDs: Lfd. Nr. 326/20
Record Dates: First submitted 2021-09-22; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Menstrual Cycle
Keywords: Immune system & metabolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — frozen EDTA and plasma samples frozen stool samples for microbial DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As there are fluctuations in the hormonal balance during the menstrual cycle, it is assumed that due to the interaction between the hormonal system and the immune system, some diseases might be worsened in the course of a cycle. This interaction is particularly important during the phases of the cycle when the corpus luteum is formed and secretes estrogens and progesterone (secretion phase, luteal phase), as well as during menstruation itself. To date, there is no comprehensive review regarding the molecular signaling pathways that are active during and influence the menstrual cycle.

The menstrual cycle influences blood glucose levels. Women are subject to greater fluctuations in blood glucose levels than men according to the phases of the menstrual cycle (menstrual phase, proliferative phase, ovulation, luteal phase). Since there are contradictory results regarding the influence of the menstrual cycle on glucose metabolism, the glucose and insulin response, as well as the glucose-dependent intestinal hormone glucagon-like peptide 1(GLP-1) after food intake are determined in the study presented here using an oral glucose tolerance test.

DETAILED DESCRIPTION:
Within the menstrual cycle there are strong hormonal fluctuations. Therefore, it is obvious that the interaction between the endocrine system and the immune system play an important role in the progression of different diseases during the course of a cycle, especially during the luteal phase and menstruation. The molecular signaling pathways that are active during the menstrual cycle and have an influence on it have not been extensively elucidated to date.

Furthermore, glucose homeostasis, on which the female cycle also can have an influence, is part of the research. Study results show that when an oral glucose tolerance test (oGTT) is performed, women are subject to greater fluctuations in blood glucose levels than men. This seems to be dependent on the phases of the female menstrual cycle. It was shown that glucose metabolism was impaired in the luteal phase. Contradictory to this, in another study no significant influence on glucose metabolism by the menstrual cycle could be detected. Based on these equivocal results, in this study the postprandial glucose and insulin response, as well of the glucose-dependent gut hormone GLP-1 in the different cycle phases will be examined.

For this purpose, an intervention study is set up in which blood samples are taken at five different time points and the subjects participate in an oGTT at four of these different time points in their individual menstrual cycle. Furthermore, anthropometry measures and body composition will be determined with the help of Bodpod and bioelectrical impedance analysis (BIA) measurements. A diary will also be kept during the entire study duration in order to record the habitual diet. In addition, different subgroups are studied: continuous measurement of body temperature or glucose levels using sensors, continuous collection of stool samples and documentation of daily nutrition using an app.

To account for regular daily variations in immunological measurements that are not related to the menstrual cycle, a cohort of healthy, male individuals will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Women or men
* Age between 20 and 30 years
* BMI: 18,5 - 25 kg/m2
* Written informed consent to participate in the study
* if applicable: Regular menstruation in the last 6 months
* if applicable: Cycle length between 21 and 35 days for each cycle in the last 6 months (self-reported).

Exclusion Criteria:

* Smoking
* Mental illness
* Chronic illnesses
* Antibiotic therapy 3 weeks before the start of the study
* Alcohol, medication and/or drug abuse (BTMG-liable or other psychotropic substances)
* Participation in another clinical study at the same time or within the last 30 days
* Hospitalization in the last 3 months
* Inflammatory condition in the last 30 days or during the course of the study
* Other exclusion criteria at the discretion of the physician/investigator
* History of infection with SARS-CoV2 before or during the study period
* Regular physical activity with very high intensity (athletes)
* Coagulation disorders
* Planning a restrictive diet for weight loss or medical reasons in the next 3 months
* Gastrointestinal disease associated with malabsorption (e.g., Crohn's disease)
* Whole blood donation within the last 3 months (women) or last 2 months (men)
* Known infertility
* Infection with Chlamydia in the past
* if applicable: Pregnancy, lactation
* if applicable: Use of any contraceptive (hormonal or chemical contraception) within and during the 6 months prior to study entry. An exception are mechanical contraceptives such as condoms
* if applicable: planning pregnancy in the next 3 months
* if applicable: attempted conception in the past 6 months
* if applicable: smear test with abnormal findings in the past 6 months (without subsequent abnormal findings)
* if applicable: untreated gynecological infection or of the urogenital tract in the last 6 months
* if applicable: gynecological surgery in the last 12 months
* if applicable: current or past other gynecologic complaints

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study participants are healthy young women with a regular menstrual cycle or heathy young men aged 20-30 years. The subjects are predominantly female students at the University of Bonn.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
characterisation of peripheral immune cells | through study completion, an average of 1 year
  scRNA-seq, PRECISE platform
gonadotropins | through study completion, an average of 1 year
  concentration of luteinizing hormone (LH), follicle stimulating hormone (FSH) (pmol/l), central laboratory, University Hospital Bonn (UKB)
sex hormones | through study completion, an average of 1 year
  concentration of estrogen, progesterone, testosterone (pmol/l), central laboratory, UKB Bonn
cytokines | through study completion, an average of 1 year
  concentration of cytokines in blood (pmol/l)

SECONDARY OUTCOMES:
glucose | during the procedure
  fasting and postprandial (after OGTT) blood glucose concentration (mg/dl), Biosen C-line, EKF
insulin | through study completion, an average of 1 year
  fasting and postprandial (after OGTT) blood insulin concentration (mU/l), central laboratory, UKB Bonn
gut microbiome | through study completion, an average of 1 year
  stool: bacterial composition of gut microbiota (diversity, taxonomy)
body height | baseline
  body height (cm), measured with stadiometer (seca scale 704, seca GmbH und Co. KG, Hamburg)
Habitual diet | baseline
  Food frequency questionnaire (FFQ), Nutrient (mg/day) and food intake (portions/day)
blood pressure | during the procedure
  blood pressure (mmHG) and heart rate (bpm), measured with Boso-carat professional, Bosch und Sohn GmbH und Co. KG, Jungingen)
body composition | during the procedure
  body composition (fat mass and fat free mass in %), measured with BIA and BOD POD
body weight | during the procedure
  body weight (kg), measured with electrical scale (seca scale 704, seca GmbH und Co. KG, Hamburg)
circumference | during the procedure
  circumference of waist and hip (cm), measure tape
GLP-1 | through study completion, an average of 1 year
  fasting and postprandial (after OGTT) blood GLP-1 concentration (pmol/l), measured by ELISA
intestinal transit time | baseline
  intestinal transit time (hours), measured by the "blue-poo" method
stool consistency | baseline
  questionnaire assessing stool consistency (Bristol-stool-scale), score from 1-7
continuous measurement of body temperature | during the procedure
  iButton (Moritz Fuchs Elektronik, Weingarten)
continuous measurement of glucose levels | during the procedure
  FreeStyle Libre 3 sensor (Abbott GmbH, Wiesbaden)
continuous collection of stool samples | during the procedure
  continuous measurement of bacterial composition of gut microbiota (diversity, taxonomy)
documentation of daily nutrition | during the procedure
  Perfood Labs App (Perfood GmbH, Lübeck), macronutrient composition (mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Rheinische Friedrich-Wilhelms-Universität Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Undecided